CLINICAL TRIAL: NCT03926377
Title: Influence of Dermocorticoids on Bone Mineral Density in Patients With Bullous Pemphigoid
Acronym: DERMOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0040
Record Dates: First submitted 2019-04-15; First posted 2019-04-24 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Osteoporosis; Bullous Pemphigoid
Keywords: osteoporosis; dermocortocoids; bullous pemphigoid; pharmacoepidemiology
MeSH Terms: conditions — Osteoporosis; Pemphigoid, Bullous | interventions — Hematologic Tests; Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clobetasol propionate treatment (Other): Clobetasol propionate (Dermoval® 0,5% cream), administered for 6 months.
  Interventions: Procedure: bone densitometry; Biological: blood test; Procedure: radiographs of the thoracic and lumbar spine; Procedure: Clobetasol propionate

INTERVENTIONS:
Procedure: bone densitometry — Patients with bullous pemphigoid will benefit from bone densitometry at the initiation of treatment, at 3 months (theoretical end of the treatment of attack) and at 6 months (theoretical end of the treatment).
Biological: blood test — Blood test of serum calcium, phosphoremia, albumin, 25 OH vitamin D and cortisol at 8 hours to highlight possible correlations between changes in bone mineral density and phosphocalcic parameters and 8 hours cortisolemia.
Procedure: radiographs of the thoracic and lumbar spine — standard radiographs of the thoracic and lumbar spine will be done at the initiation of treatment and at 6 months.
Procedure: Clobetasol propionate — Clobetasol propionate (Dermoval® 0,5% cream), administered for 6 months.

SUMMARY:
Bullous pemphigoid is the most common type of bullous skin disease and is clinically characterized by clear-tense bullae, which result in post-bullous cutaneous erosions, altering the skin barrier. The treatment of this pathology consists of the application of high doses of topical corticosteroids (clobetasol propionate) for a prolonged period of at least 6 months. The main objective of this study is to demonstrate a change in bone mineral density at 6 months after initiation of treatment, in subjects with bullous pemphigoid and treated with topical corticosteroid.

DETAILED DESCRIPTION:
Glucocorticoids have direct effects on bone remodeling by suppressing bone formation (inhibition of osteoblastic differentiation, inhibition of mature osteoblasts function and apoptosis of mature osteoblasts) and by increasing bone resorption (decrease in osteoclast apoptosis and stimulation of osteoclastogenesis). They also have indirect bone effects by decreasing the intestinal absorption of calcium and increasing its urinary excretion, and by inhibiting the somatotropic and gonadotropic axis. This pathophysiology results in excessive bone fragility. Bone loss and increased incidence of fractures occur within 6 months after the introduction of oral corticosteroid therapy, with a partially reversible phenomenon within months of discontinuation. The extent of bone loss depends on the dose and duration of glucocorticoid administration.

The systemic transition of topical corticosteroids depends on several parameters such as excipients, anatomical location, cutaneous state, the dose used and the duration of exposure.

Clobetasol propionate, used for long-term use in bullous pemphigoid, is a Class IV dermocorticoid (highly potent). Patients with bullous pemphigoid will benefit from bone densitometry at the initiation of treatment, at 3 months (theoretical end of the treatment of attack) and at 6 months (theoretical end of the treatment).

Patients will also benefit a blood test of serum calcium, phosphoremia, albumin, 25 OH vitamin D and cortisol at 8 to highlight possible correlations between changes in bone mineral density and phosphocalcic parameters and 8 cortisolemia (braking of the hypothalamic-pituitary-adrenal axis).

Patients will also benefit from standard radiographs of the thoracic and lumbar spine at the initiation of treatment and at 6 months. Follow-up is planned over 6 months, with 2 follow-up visits at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting a multi-bullous pemphigoid newly diagnosed or relapsed more than 3 months after stopping corticosteroids and treated according to the national protocol for diagnosis and care issued by the reference center for autoimmune bullous diseases of April 2016
* patients having received written and oral information and signed informed consent
* patients covered by national health insurance

Exclusion Criteria:

* Patients under tutorship or curatorship or inability to give informed consent
* Patients receiving an anti-osteoporotic treatment
* Patients requiring an anti-osteoporotic baseline treatment (T-score ⩽ -3DS on at least 1 site or FRAX score above the therapeutic intervention threshold)
* Patients with one or more major risk factors for osteoporosis
* Patients who have received topical corticosteroids in less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Variation of the bone mineral density (BMD) expressed in g/cm² at the lumbar spine between baseline and the theorical end of the treatment. | 6 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from bone densitometry at the initiation of the treatment and at 6 months (theoretical end of the treatment).

SECONDARY OUTCOMES:
Variation of the bone mineral density (BMD) expressed in g/cm² at the lumbar spine between baseline and the theorical end of the treatment of attack. | 3 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from bone densitometry at the initiation of the treatment and at 3 months (theoretical end of the treatment of attack).
Variation of the bone mineral density (BMD) expressed in g/cm² at the hip between baseline and the theorical end of the treatment of attack. | 3 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from bone densitometry at the hip at the initiation of the treatment and at 3 months (theoretical end of the treatment of attack).
Variation of the bone mineral density (BMD) expressed in g/cm² at the hip between baseline and the theorical end of the treatment. | 6 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from bone densitometry at the hip at the initiation of the treatment and at 6 months (theoretical end of the treatment).
Variation in plasma concentrations of corrected calcemia, phosphoremia, 25 OH vitamin D and cortisolemia between Baseline and the theorical end of the treatment of attack. | 3 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from a blood test of serum calcium, phosphoremia, albumin, 25 OH vitamin D and cortisol at 8h at the initiation of the treatment and at 3 months (theoretical end of the treatment attack).
Variation in plasma concentrations of corrected calcemia, phosphoremia, 25 OH vitamin D and cortisolemia between Baseline and the theorical end of the treatment. | 6 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from a blood test of serum calcium, phosphoremia, albumin, 25 OH vitamin D and cortisol at 8h at the initiation of the treatment and at 6 months (theoretical end of the treatment).
frequency of fractures (axial and , or peripheral) | 6 months after beginning of the treatment
  Patients with bullous pemphigoid and treated with Clobetasol propionate will benefit from standard radiographs of the thoracic and lumbar spine at the initiation of the treatment and at 6 months (theoretical end of the treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Chaby, MD, Principal Investigator — CHU Amiens; Catherine Lok, Pr, Principal Investigator — CHU Amiens; Pascal Joly, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No